CLINICAL TRIAL: NCT01794572
Title: Phase 1-2 Study of the Combination of Escalated Total Bone Marrow Irradiation (TBMI) by Helicoidal Tomotherapy and a Fixed High-dose Melphalan (140 mg/m²) Followed by Peripheral Stem Cell Rescue (PSC) in First Relapsed Multiple Myeloma.
Brief Title: Phase 1-2 Study of Total Bone Marrow Irradiation With Helicoidal Tomotherapy in 1st Myeloma Relapse
Acronym: TOMMY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient recruitement rate and modification of the therapeutic standard
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-2012-04; 2012-001473-91 (EudraCT Number)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; Relapse; Complete Remission; Very Good Partial Remission
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: Total Bone Marrow Irradiation (TBMI) dose escalation
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Total Bone Marrow Irradiation (TBMI): 8 Gy (Experimental): Cohort 1: Total Bone Marrow Irradiation (TBMI): 8 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
  Interventions: Radiation: Total Bone Marrow Irradiation (TBMI) 8 Gy
- Total Bone Marrow Irradiation (TBMI): 10 Gy (Experimental): Cohort 2: Total Bone Marrow Irradiation (TBMI): 10 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
  Interventions: Radiation: Total Bone Marrow Irradiation (TBMI) 10 Gy
- Total Bone Marrow Irradiation (TBMI): 12 Gy (Experimental): Cohort 3: Total Bone Marrow Irradiation (TBMI): 12 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
  Interventions: Radiation: Total Bone Marrow Irradiation (TBMI): 12 Gy
- Cohort 4: Total Bone Marrow Irradiation (TBMI): 14 Gy (Experimental): Cohort 4: Total Bone Marrow Irradiation (TBMI): 14 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
  Interventions: Radiation: Total Bone Marrow Irradiation (TBMI): 14 Gy
- Total Bone Marrow Irradiation (TBMI): 16 Gy (Experimental): Cohort 5: Total Bone Marrow Irradiation (TBMI): 16 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
  Interventions: Radiation: Total Bone Marrow Irradiation (TBMI): 16 Gy

INTERVENTIONS:
Radiation: Total Bone Marrow Irradiation (TBMI) 8 Gy — Total Bone Marrow Irradiation (TBMI): 8 Gy
  Arms: Total Bone Marrow Irradiation (TBMI): 8 Gy
Radiation: Total Bone Marrow Irradiation (TBMI) 10 Gy — Total Bone Marrow Irradiation (TBMI): 10 Gy
  Arms: Total Bone Marrow Irradiation (TBMI): 10 Gy
Radiation: Total Bone Marrow Irradiation (TBMI): 12 Gy — Total Bone Marrow Irradiation (TBMI): 12 Gy
  Arms: Total Bone Marrow Irradiation (TBMI): 12 Gy
Radiation: Total Bone Marrow Irradiation (TBMI): 14 Gy — Total Bone Marrow Irradiation (TBMI): 14 Gy
  Arms: Cohort 4: Total Bone Marrow Irradiation (TBMI): 14 Gy
Radiation: Total Bone Marrow Irradiation (TBMI): 16 Gy — Total Bone Marrow Irradiation (TBMI): 16 Gy
  Arms: Total Bone Marrow Irradiation (TBMI): 16 Gy

SUMMARY:
In Multiple Myeloma, an adult hematological malignancy, mainly located in the Bone Marrow (BM), dramatic recent progresses have been observed, thanks to new agents (proteasome inhibitors and IMIDs). However, at time of first relapse, high-dose therapy followed by Stem Cell Rescue (SCR) is frequently mandatory as a consolidation in minimal residual disease, to healthy patients under 65 yo, combining Melphalan (MPH) and/or Total Body Irradiation. Modern irradiation modalities are now available by the use of HI-ART Tomotherapy system to realize a Total Bone Marrow Irradiation (TBMI), in order both to limit the dose administered to Organ at Risk (lungs, oral cavity) and to focus efficacy on BM. In this phase-1 study, the conditioning regimen before SCR will combine a fixed high-dose MPH (140 mg/m²) and a dose escalated TBMI, so as to define its Maximal Tolerated Dose (MTD) and the Dose Limiting Toxicities (DLT). An extended cohort will further in a phase-2 setting.

DETAILED DESCRIPTION:
Experimental :

Total Bone Marrow Irradiation (TBMI) is delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3. The escalated dose levels are determined according to a "3x3" modified Fibonacci method and five dose levels will be explored. The doses per fraction are: 1gy, 1.25gy, 1.5gy, 1.75gy and 2gy, and consequently the cumulative TBMI doses are: 8gy, 10gy, 12gy, 14gy and 16gy.

Drug : Melphalan is infused intravenously in 30 minutes on day -2 after IV anti-emetics.

Autologous Peripheral Stem Cell Rescue : are re-infused in the central line on day "0" after adequate premedication.

Despite the recent finding of new drugs (proteasome inhibitors and IMIDs), Multiple Myeloma still remain uncurable, especially after the first relapse, even in responding disease under conventional chemotherapy. In the healthy youngest patients (<65 yo), when peripheral stem cells collection is available, a high-dose therapy is often proposed in consolidation of complete or very good partial remission: the conditioning regimen usually includes high dose alkylating agent (mostly Melphalan) and/or Total Body Irradiation. The new Tomotherapy HI-ART technology allows irradiating on a 1.6m length field all the bone marrow sites together with optimal respect of the Organ at Risk (lungs, oral cavity, heart, liver, kidneys…). The proposed phase-1 study will explore the safety and efficacy of escalated dose of Total Bone-Marrow Irradiation in combination with a fixed dose of Melphalan (140mg/m²), followed by autologous SCR. To determine the MTD is the main objective of the study, then the toxicity profile (DLTs) and the RP2D in an extended cohort at the MTD dose.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma in first relapse.
* In Complete or very good partial remission
* Available Collected Autologous Peripheral Stem cells: 2.5x106 CD34+/Kg

Exclusion Criteria:

* Uncontrolled visceral disease: kidney, heart, lung, diabetes mellitus
* Previous Total body irradiation
* Any previous radiation dose to the spinal cord which could reach to 45gy equivalent, including the proposed TBMI
* Amyloidosis
* Brain localizations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane A SUPIOT, MD, PhD, Principal Investigator — Institut de Cancerologie de l'Ouest; Philippe MOREAU, MD, PhD, Principal Investigator — University Hospital, CHU de NANTES
Locations (8):
- France (8):
  - CLCC Bergonie, service de radiotherapie, Bordeaux
  - CHU Haut-Leveque, service d'Hématologie, Bordeaux
  - CLCC Oscar Lambret, service de radiothérapie, Lille
  - CHU Claude Huriez, service d'hématologie, Lille
  - CHU Hotel-Dieu, service d'hématologie, Nantes
  - CLCC ICO, service de radiothérapie, Saint-Herblain
  - CLCC Paul Strauss, service de radiothérapie, Strasbourg
  - CHU Hautepierre, service d'hématologie, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong JY, Rosenthal J, Liu A, Schultheiss T, Forman S, Somlo G. Image-guided total-marrow irradiation using helical tomotherapy in patients with multiple myeloma and acute leukemia undergoing hematopoietic cell transplantation. Int J Radiat Oncol Biol Phys. 2009 Jan 1;73(1):273-9. doi: 10.1016/j.ijrobp.2008.04.071. Epub 2008 Sep 9. PMID 18786784
- [Background] Somlo G, Spielberger R, Frankel P, Karanes C, Krishnan A, Parker P, Popplewell L, Sahebi F, Kogut N, Snyder D, Liu A, Schultheiss T, Forman S, Wong JY. Total marrow irradiation: a new ablative regimen as part of tandem autologous stem cell transplantation for patients with multiple myeloma. Clin Cancer Res. 2011 Jan 1;17(1):174-82. doi: 10.1158/1078-0432.CCR-10-1912. Epub 2010 Nov 3. PMID 21047977
- See also: Publication in International journal of radiation oncology . biology . physics — https://doi.org/10.1016/j.ijrobp.2022.09.069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: April 9, 2013 Study completion date: October 6, 2020
Groups:
- Total Bone Marrow Irradiation (TBMI): 10 Gy: Cohort 1: Total Bone Marrow Irradiation (TBMI): 10 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
- Total Bone Marrow Irradiation (TBMI): 14 Gy: Cohort 4: Total Bone Marrow Irradiation (TBMI): 14 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue : re-infused in the central line on day "0" after adequate premedication.
Period: Overall Study
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy
Started | 3 | 3 | 6 | 1 | 0
Completed | 3 | 3 | 6 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated prematurely, due to a lack of enrolments
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy | Total
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6 | 1 | 0 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 1 | 0 | 5
  Male | 3 | 1 | 4 | 0 | 0 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  France | 3 | 3 | 6 | 1 |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose, Type of DLTs
Description: Maximal Tolerated Dose Type of Dose-limiting Toxicities The escalated dose levels are determined according to a "3x3" modified Fibonacci method and five dose levels will be explored. The doses per fraction are: 1gy, 1.25gy, 1.5gy, 1.75gy and 2gy, and consequently the cumulative TBMI doses are: 8gy, 10gy, 12gy, 14gy and 16gy.
Time Frame: 1 year
Population: The study was terminated prematurely, due to a lack of enrolments
Measure: Count of Participants; unit: Participants
Groups:
- Total Bone Marrow Irradiation (TBMI): 10 Gy: Cohort 2: Total Bone Marrow Irradiation (TBMI): 10 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue: re-infused in the central line on day "0" after adequate premedication.
- Total Bone Marrow Irradiation (TBMI): 12 Gy: Cohort 3: Total Bone Marrow Irradiation (TBMI): 12 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue: re-infused in the central line on day "0" after adequate premedication.
- Total Bone Marrow Irradiation (TBMI): 14 Gy: Cohort 4: Total Bone Marrow Irradiation (TBMI): 14 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue: re-infused in the central line on day "0" after adequate premedication.
- Total Bone Marrow Irradiation (TBMI): 16 Gy: Cohort 5: Total Bone Marrow Irradiation (TBMI): 16 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue: re-infused in the central line on day "0" after adequate premedication.
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 0
Participants
  DLT: Severe sepsis | 0 | 0 | 1 | 0 |
  Patients without DLT | 3 | 3 | 5 | 1 |

2. Secondary Outcome: Safety Profile Recommended Dose for Phase-2 (RDP2)
Description: Safety profile: acute, short and middle term toxicities Recommended Dose for Phase-2 (RDP2) and Extended Cohort for 14 patients at this dose
Time Frame: 1 year
Population: The study was terminated prematurely, due to a lack of enrolments. The recommended dose for phase-2 has not been reached. No extended cohort has been performed
Measure: Count of Participants; unit: Participants
Groups:
- Total Bone Marrow Irradiation (TBMI): 8 Gy: Cohort 1: Total Bone Marrow Irradiation (TBMI): 8 Gy delivered by the Tomotherapy HI-ART machine, in 2 fractions per day during 4 consecutive days from d -6 to d -3.
  Melphalan 140 mg/m² infused intravenously during 30 minutes on day -2 after IV anti-emetics.
  Autologous Peripheral Stem Cell Rescue: re-infused in the central line on day "0" after adequate premedication.
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 0
Participants
  Recommended dose reached | 0 | 0 | 0 | 0 | 0
  Patients treated at lower dose levels | 3 | 3 | 6 | 1 |
  Extended Cohort performed | 0 | 0 | 0 | 0 |

3. Other Pre Specified Outcome: Efficacy Expressed as the Rate (%) of Complete Response and Very Good Partial Response
Description: osteo-medullary PET fixations evaluation by FDG PET-Scan Disease-free survival at 1 year and Overall Survival
Time Frame: 1 and 2 years
Population: The study was terminated prematurely, due to a lack of enrolments
Measure: Count of Participants; unit: Participants
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 0
Participants
  Patients with very good partial response | 1 | 1 | 3 | 0 |
  Patients with partial response | 2 | 0 | 2 | 0 |
  Patients with complete response | 0 | 2 | 1 | 1 |

ADVERSE EVENTS:
Time Frame: The adverse events were collected from enrollment until 90 days post Autologous Peripheral Stem Cell (PSC) Rescue.
Description: The study was terminated prematurely, due to a lack of enrolments. All Serious adverse events, adverse events and all-cause mortality are reported.
Arm/Group | Total Bone Marrow Irradiation (TBMI): 8 Gy | Total Bone Marrow Irradiation (TBMI): 10 Gy | Total Bone Marrow Irradiation (TBMI): 12 Gy | Total Bone Marrow Irradiation (TBMI): 14 Gy | Total Bone Marrow Irradiation (TBMI): 16 Gy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/6 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Bone Marrow Irradiation (TBMI): 8 Gy (N=3) | Total Bone Marrow Irradiation (TBMI): 10 Gy (N=3) | Total Bone Marrow Irradiation (TBMI): 12 Gy (N=6) | Total Bone Marrow Irradiation (TBMI): 14 Gy (N=1) | Total Bone Marrow Irradiation (TBMI): 16 Gy (N=0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Acute Grade 3 diarrhoea related to Melphalan
Dyspnoea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dyspnoea grade 3 related to anemia
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Septic shock grade 3 with febrile neutropenia
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Implanted-port-catheter-related sepsis caused by Staphylococcus aureus grade 3
Severe cognitive distress (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Severe cognitive distress associated to hypernatremia and febrile aplasia grade 3
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Febrile episode consistent with engraftment syndrome following stem cell transplantation, grade 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Interstitial lung disease with cytokine release syndrome grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Bone Marrow Irradiation (TBMI): 8 Gy (N=3) | Total Bone Marrow Irradiation (TBMI): 10 Gy (N=3) | Total Bone Marrow Irradiation (TBMI): 12 Gy (N=6) | Total Bone Marrow Irradiation (TBMI): 14 Gy (N=1) | Total Bone Marrow Irradiation (TBMI): 16 Gy (N=0)
Thrombopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 6 (8) | 1 (1) | NA — Grade 3 and 4
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA — Sepsis due to Staphylococcus hominis, grade 3
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 4 (5) | 1 (1) | NA — Grade 3 to 4
Mucositis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | NA — Grade 3 to 4
Febrile aplasia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 3 to 4
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | NA — Grade 3
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 3
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 3
Hypocalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 4
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 3
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | NA — Grade 3 to 4
Leucopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | NA — Grade 3 to 4
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | NA — Grade 2
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA — Grade 2
Thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA — Grade 2
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA — Grade 2
Neuropathic flare-up (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA — Grade 2
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA — Grade 2
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA — Grade 2
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA — Grade 1
Radiodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 1
Streptococcus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 2
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 1
Lower limb edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT01794572/Prot_SAP_000.pdf